CLINICAL TRIAL: NCT02606175
Title: Medication Knowledge, Medication Adherence and Health Literacy in Patients Who Underwent a Kidney Transplantation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: s58561
Record Dates: First submitted 2015-10-27; First posted 2015-11-17 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2018-10

CONDITIONS: Adherence to Medication Regime
Keywords: health literacy; patient medication knowledge; kidney transplantation; medication adherence; kidney transplant; renal transplantation
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Admitted for renal transplantation (Other): Patients who are hospitalised on the abdominal transplantation surgery ward at the University Hospitals of Leuven (UZLeuven) and undergo a kidney transplantation during this hospitalisation.
  Intervention: taking questionnaires and tests at predefined timepoints:
  * at discharge: NVS-D, FCCHL, BAASIS, medication knowledge test, demographic factors questionnaire
  * 1 month after kidney transplantation: BAASIS, medication knowledge test
  * 3 months after kidney transplantation: NVS-D, FCCHL, BAASIS, medication knowledge test
  * 1 year after kidney transplantation: NVS-D, FCCHL, BAASIS, medication knowledge test, demographic factors questionnaire
  * 2 years after kidney transplantation: NVS-D, FCCHL, BAASIS, medication knowledge test, demographic factors questionnaire
  Interventions: Other: Taking questionnaires and tests

INTERVENTIONS:
Other: Taking questionnaires and tests — At predefined timepoints:
  * 2 tests for health literacy: New Vital Sign-Dutch version (NVS-D) and Functional, Communicative and Critical Health Literacy (FCCHL)
  * 1 test for medication adherence: BAASIS
  * 1 questionnaire about demographic factors (weight, income, sex, age, financial situation,...)
  * 1 test about medication knowledge

SUMMARY:
Patients who receive a kidney transplant have to learn in 10-14 days which anti-rejection medication to take, how to take it ,... This learning process is attended by the nurses of the ward. This study wants to measure the degree of medication knowledge, health literacy and medication adherence of those patients.

DETAILED DESCRIPTION:
Patients who receive a kidney transplant arrive at the abdominal transplantation surgery ward after surgery. Within 10-14 days they learn which anti-rejection medication they have to take, how they have to take it and to what they have to pay attention. This learning process is attended by the nurses of the ward.

It is already known that a bad medication adherence is related to a higher rejection rate and mortality of patients who receive a kidney transplant. Bad medication knowledge and low health literacy are correlated with a bad medication adherence. Data about the level of health literacy of the Belgian population (and certainly of patients who just received a kidney transplant) are scarce.

The main purpose of this study is to have an idea of the extent of medication knowledge, heath literacy and adherence in patients who received a renal transplant.

Therefore, a prospective cohort study will be performed. Adult patients admitted for a renal transplantation, will be included after obtainment of informed consent. The patients will be followed for 2 years. On predefined time points, the participants will have to fill in questionnaires and tests: on discharge 2 tests that measure health literacy, the "Basel Assessment of Adherence to Immunosuppressive Medications Scale" (BAASIS), the medication knowledge test and a questionnaire about demographic factors. At 1 month post-transplantation the BAASIS test and medication knowledge test, 3 months post-transplantation the 2 tests assessing health literacy, the BAASIS test and medication knowledge test and finally after 1 and 2 years all the tests (4 in total) and questionnaire assessing demographic factors

ELIGIBILITY:
Inclusion Criteria: patients who are admitted at the abdominal transplantation surgery ward and just underwent a kidney transplantation

Exclusion Criteria:

* Patients who cannot sufficiently write, read or speak Dutch.
* Patients who don't take care of their medication themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Degree of medication knowledge pre-and post kidney transplantation as measured by the self-edited medication knowledge test | Up to 36 months
  Measurement: quantitative score
Degree of health literacy pre- and post kidney transplantation as measured by the NVS-D and FCCHL test | Up to 36 months
  Measurement: NVS-D = quantitative score (max = 6 points) with 3 groups: low health literacy = 0-1; intermediate health literacy = 2-3; high health literacy = 4-6.
  The FCCHL contains 3 subitems (functional, communicative and critical health literacy) Each subitem contains 4 questions. Each question is rated on a 4-point scale, ranging from 1 to 4 (4 indicating high health literacy). The scores for the items in a scale are summed and divided by the number of items in the scale to give a scale score (theoretical range 1-4).
Degree of medication adherence pre- and post kidney transplantation assessed by the BAASIS test | Up to 36 months
  Measurement: BAASIS = 4 questions assessing adherence. If the patient answers 'no' on at least 1 question, the patient is categorized as 'non-adherent'.

SECONDARY OUTCOMES:
Type of evolution in the degree of medication knowledge (assessed by self-edited test, see above), health literacy (assessed by NVS-D and FCCHL, see above) and/or medication adherence (assessed by BAASIS, see above). | Up to 36 months
  Is their a positive or negative evolution in medication knowledge, health literacy and/or medication adherence at discharge-1month-3 months-1 year-2 years after kidney transplantation?
Correlation between degree of medication knowledge, degree of health literacy and/or degree of medication adherence | Up to 36 months
Correlation between evolution of medication knowledge, evolution of health literacy and/or evolution of medication adherence | Up to 36 months
Defining risk factors (assessed by the demographic questionnaire) related to the degree of medication knowledge, health literacy and/or medication adherence | Up to 36 months
Defining risk factors (assessed by the demographic questionnaire) related to the evolution of medication knowledge, health literacy and/or medication adherence | Up to 36 months
Correlation between the degree of medication knowledge, health literacy and/or medication adherence, and outcome parameters (trend of serum creatinine, result of biopsy of kidney transplant, trend and variation of tacrolimus' trough level) | Up to 36 months
Correlation between the evolution of medication knowledge, health literacy and/or medication adherence, and the outcome parameters (trend of serum creatinine, result of biopsy of kidney transplant, trend and variation of tacrolimus' trough level). | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Adams, Principal Investigator — UZ Leuven; Barbara Deleenheer, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hartono C, Muthukumar T, Suthanthiran M. Immunosuppressive drug therapy. Cold Spring Harb Perspect Med. 2013 Sep 1;3(9):a015487. doi: 10.1101/cshperspect.a015487. PMID 24003247
- [Background] Pinsky BW, Takemoto SK, Lentine KL, Burroughs TE, Schnitzler MA, Salvalaggio PR. Transplant outcomes and economic costs associated with patient noncompliance to immunosuppression. Am J Transplant. 2009 Nov;9(11):2597-606. doi: 10.1111/j.1600-6143.2009.02798.x. PMID 19843035
- [Background] Vlaminck H, Maes B, Evers G, Verbeke G, Lerut E, Van Damme B, Vanrenterghem Y. Prospective study on late consequences of subclinical non-compliance with immunosuppressive therapy in renal transplant patients. Am J Transplant. 2004 Sep;4(9):1509-13. doi: 10.1111/j.1600-6143.2004.00537.x. PMID 15307839
- [Background] Ponticelli C, Graziani G. Education and counseling of renal transplant recipients. J Nephrol. 2012 Nov-Dec;25(6):879-89. doi: 10.5301/jn.5000227. PMID 23042431
- [Background] LaFleur J, Oderda GM. Methods to measure patient compliance with medication regimens. J Pain Palliat Care Pharmacother. 2004;18(3):81-7. PMID 15364635
- [Background] Dobbels F, Berben L, De Geest S, Drent G, Lennerling A, Whittaker C, Kugler C; Transplant360 Task Force. The psychometric properties and practicability of self-report instruments to identify medication nonadherence in adult transplant patients: a systematic review. Transplantation. 2010 Jul 27;90(2):205-19. doi: 10.1097/TP.0b013e3181e346cd. PMID 20531073
- [Background] De Geest S, Borgermans L, Gemoets H, Abraham I, Vlaminck H, Evers G, Vanrenterghem Y. Incidence, determinants, and consequences of subclinical noncompliance with immunosuppressive therapy in renal transplant recipients. Transplantation. 1995 Feb 15;59(3):340-7. PMID 7871562
- [Background] Zhang NJ, Terry A, McHorney CA. Impact of health literacy on medication adherence: a systematic review and meta-analysis. Ann Pharmacother. 2014 Jun;48(6):741-51. doi: 10.1177/1060028014526562. Epub 2014 Mar 11. PMID 24619949
- [Background] Sorensen K, Van den Broucke S, Fullam J, Doyle G, Pelikan J, Slonska Z, Brand H; (HLS-EU) Consortium Health Literacy Project European. Health literacy and public health: a systematic review and integration of definitions and models. BMC Public Health. 2012 Jan 25;12:80. doi: 10.1186/1471-2458-12-80. PMID 22276600
- [Background] Fransen MP, Leenaars KE, Rowlands G, Weiss BD, Maat HP, Essink-Bot ML. International application of health literacy measures: adaptation and validation of the newest vital sign in The Netherlands. Patient Educ Couns. 2014 Dec;97(3):403-9. doi: 10.1016/j.pec.2014.08.017. Epub 2014 Sep 3. PMID 25224314
- [Background] van der Vaart R, Drossaert CH, Taal E, ten Klooster PM, Hilderink-Koertshuis RT, Klaase JM, van de Laar MA. Validation of the Dutch functional, communicative and critical health literacy scales. Patient Educ Couns. 2012 Oct;89(1):82-8. doi: 10.1016/j.pec.2012.07.014. Epub 2012 Aug 9. PMID 22878030
- [Background] Heijmans M, Waverijn G, Rademakers J, van der Vaart R, Rijken M. Functional, communicative and critical health literacy of chronic disease patients and their importance for self-management. Patient Educ Couns. 2015 Jan;98(1):41-8. doi: 10.1016/j.pec.2014.10.006. Epub 2014 Oct 16. PMID 25455794